CLINICAL TRIAL: NCT02950974
Title: Change in Serum Chloride Level After Loading Dose of Sterofundin Solution Compared With Normal Saline Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Cherdkiat karnjanarachata, Dr., Ramathibodi Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Stero
Record Dates: First submitted 2016-10-27; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Change in Serum Chloride Level
Keywords: sterofundin; resuscitation; normal saline; chloride; fluid; SID; pH; osmolality; urine
MeSH Terms: conditions — Sudden Infant Death | interventions — sterofundin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NSS (Active Comparator): NSS 30 ml/kg (maximum of 2 litres) intravenous load over 1 hour
  Interventions: Drug: Sterofundin; Drug: NSS
- Sterofundin (Experimental): Sterofundin solution 30 ml/kg (maximum of 2 litres) intravenous load over 1 hour
  Interventions: Drug: Sterofundin; Drug: NSS

INTERVENTIONS:
Drug: Sterofundin — Fluid loading
Drug: NSS — Fluid loading

SUMMARY:
Prospective, crossover, randomized trial to evaluate plasma compositions after loading dose of sterofundin solution given to healthy volunteer in the resuscitation manner compared with normal saline solution.

DETAILED DESCRIPTION:
10 healthy volunteers were randomly assigned to receive either normal saline or sterofundin for the first solution in dose of 30 mL/kg (max 2 L) over 1 hour. Blood was collected at baseline (T0), at 60 minutes (T1), 120 minutes (T2), and 240 minutes (T4) from baseline. Time to fist void after initiation of fluid and urine volume were also recorded. After wash-out period of at least 1 week, crossover studies were performed with another fluid.

ELIGIBILITY:
Inclusion Criteria:

* No underlying disease
* LVEF > 0.5
* No current medication usage

Exclusion Criteria:

* Pregnancy or lactation
* BMI <18 or >25
* Fever presented in the past 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in serum chloride | 4 hours
  At 0, 1, 2, and 4 hours from initiation

SECONDARY OUTCOMES:
Change in serum pH | 4 hours
  At 0, 1, 2, and 4 hours from initiation
Change in serum osmolality | 4 hours
  At 0, 1, 2, and 4 hours from initiation
Change in serum SID | 4 hours
  At 0, 1, 2, and 4 hours from initiation
Time to first void | Within 24 hours
  Time in minutes from initiation of fluid to first urination
Urine volume | Within 24 hours
  Volume of first urination in ml

CONTACTS AND LOCATIONS:
Overall Officials: Sunthiti Morakul, MD, Principal Investigator — Ramathibodi Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awad S, Allison SP, Lobo DN. The history of 0.9% saline. Clin Nutr. 2008 Apr;27(2):179-88. doi: 10.1016/j.clnu.2008.01.008. Epub 2008 Mar 3. PMID 18313809
- [Background] Chowdhury AH, Cox EF, Francis ST, Lobo DN. A randomized, controlled, double-blind crossover study on the effects of 2-L infusions of 0.9% saline and plasma-lyte(R) 148 on renal blood flow velocity and renal cortical tissue perfusion in healthy volunteers. Ann Surg. 2012 Jul;256(1):18-24. doi: 10.1097/SLA.0b013e318256be72. PMID 22580944
- [Background] Yunos NM, Bellomo R, Hegarty C, Story D, Ho L, Bailey M. Association between a chloride-liberal vs chloride-restrictive intravenous fluid administration strategy and kidney injury in critically ill adults. JAMA. 2012 Oct 17;308(15):1566-72. doi: 10.1001/jama.2012.13356. PMID 23073953
- [Background] Morgan TJ, Venkatesh B, Hall J. Crystalloid strong ion difference determines metabolic acid-base change during acute normovolaemic haemodilution. Intensive Care Med. 2004 Jul;30(7):1432-7. doi: 10.1007/s00134-004-2176-x. Epub 2004 Feb 28. PMID 14991093